CLINICAL TRIAL: NCT07024329
Title: Implementing REmote SymPtom mOnitoring and maNagement (RESPONd): Evaluating the Impact on Cancer Patients, System Efficiency, and Economic Outcomes
Brief Title: Implementing REmote SymPtom mOnitoring and maNagement (RESPONd)
Acronym: RESPONd
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other); Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Linda Watson, Executive Director, Supportive Care Services and Patient Experience, Cancer Care Alberta, Alberta Health Services, University of Calgary
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HREBA.CC-24-0138
Record Dates: First submitted 2025-05-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Patient Reported Outcomes; Quality of Life; Clinical Decision Making; Patient Reported Outcome Measures; Patient Experience; Health Service Utilization; Symptom Management; PROMs; PROs
MeSH Terms: conditions — Neoplasms; Patient Acceptance of Health Care | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESPONd (Experimental): Participants will be recruited and supported to complete electronic PROs questionnaires. Study nurses will monitor the electronic PROs completed between clinic visits and contact patients to provide personalized support.
  Interventions: Other: Remote Symptom Monitoring and Management; Other: Clinic Team Huddle
- Non-RESPONd (No Intervention): Usual care.

INTERVENTIONS:
Other: Remote Symptom Monitoring and Management — A study nurse will digitally monitor symptom complexity and provide symptom management between clinic visits. This will increase the frequency of collection and use of electronic PROs to provide responsive symptom management. Electronic PROs are collected digitally, and a complexity algorithm is used to flag patients with high symptom complexity. This will allow the study nurse to proactively manage symptoms in a timelier way.
  Arms: RESPONd
Other: Clinic Team Huddle — Support will be provided to clinic teams to implement a team huddle (team planning session) one week prior to clinics, to assess how additional electronic PROs data for patients participating in RESPONd impacts their ability to identify stable patients with low symptom complexity who could receive virtual care or Registered Nurse (RN) led clinic care.
  Arms: RESPONd

SUMMARY:
The goal of this study is to understand if the implementation of a remote symptom monitoring and management program improves outcomes. The program will provide patients the opportunity to complete electronic Patient Reported Outcomes (PROs) questionnaires from home between appointments and receive tailored advice from a study nurse. A second goal of this study is to examine the impact of electronic symptom monitoring on clinic efficiencies.

The main question it aims to answer is:

• What impact does implementing digitally enabled remote symptom monitoring and management (RESPONd) between ambulatory oncology visits have on patient outcomes and system efficiencies?

Participants will:

* Report their symptoms and concerns from home by completing the electronic symptom monitoring questionnaire.
* Discuss their symptoms and concerns with a study nurse.
* Provide feedback about their experience at important timepoints during the study.
* Participate as usual in ambulatory clinic appointments.

DETAILED DESCRIPTION:
Rationale:

In recent years, cancer care has increasingly shifted from acute to ambulatory settings as a strategy to manage healthcare costs. While some emergency department (ED) visits are unavoidable due to the complexity of cancer-related issues, many could be prevented through timely symptom management and coordinated care in ambulatory oncology. The integration of Patient Reported Outcomes (PROs) into routine cancer care has been shown to reduce ED visits, enhance quality of life, and improve overall survival.

Within Cancer Care Alberta, PROs are routinely collected during clinic visits and electronically, using a standardized questionnaire that assesses common symptoms and supportive care needs experienced by cancer patients. Despite this, the use of electronic PROs data for real-time symptom management remains inconsistent, and there is currently no established workflow in Alberta for remote symptom monitoring. As a result, healthcare providers often lack advance insight into patients' symptoms prior to appointments.

Study Design:

The study is a stepped-wedge effectiveness-implementation type 1 hybrid design. RESPONd will be implemented over 1.5 years in six clinics, spanning tertiary, regional, and community cancer centres. Study nurses will monitor electronic PROs questionnaires completed between clinic visits and contact patients to provide personalized support. Collected electronic PROs information will also be utilized during weekly triage discussions in each clinic, where the route of care will be tailored for patients based on their symptom complexity. Participant quality of life will be measured at baseline, 3, and 6 months. Health care utilization compared to non-RESPONd patients will be evaluated. The implementation of this study will be evaluated using the RE-AIM framework, utilizing all constructs.

Potential impact on practice:

The study will explore a person-centered, proactive approach to remote symptom management and the effects on patient experience, outcomes, and clinical teams. RESPONd represents an innovative opportunity to shift the model of care in oncology clinics to optimize efficiency and utilization of limited clinic resources and create a responsive care team that is ready and able to provide personalized symptom management and supportive care within the cancer journey.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Have cancer
* Receiving care in one of the participating clinics.
* Able to sign up for MyAHS Connect and consent.
* Have access to a digital device at home
* Able to complete their electronic PROs questionnaire without support from the clinic team on a weekly (patients on active treatment) or monthly (patients on follow-up) basis, for the duration of the intervention or until they are discharged from the clinic.
* Regular access to a telephone in order for the study nurse to call patients to provide symptom management support.

Exclusion Criteria:

* Patients with cognitive disabilities or who cannot reliably report symptoms independently.
* Patients not residing in Alberta, as government-issued ID is required to register for MyAHS Connect.
* Patients who do not have regular access to a telephone, as the study nurse needs to be able to call patients to provide symptom management support.
* Patients who do not speak English, or who do not have an English-speaking friend, family member, or caregiver to assist them, as the electronic PROs questionnaire is only available in English at this time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1055 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL) | Baseline, 3 months and 6 months
  RESPONd participants will be asked to complete the Euro Quality of Life -EuroQol-5 Dimension 5 Level (EQ-5D-5L) questionnaire. This is a generic measure of QoL often used with cancer patients. Consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with 5 levels (from no problems to extreme problems).
  The responses form a 5-digit health state profile (e.g., 11111 = perfect health).
  These profiles are converted into a single summary index value (utility score) using a Canadian-specific value set derived through the Time Trade-Off (TTO) method.
  Utility Index Score Range (Canada):
  Minimum: Less than 0 (indicating a health state considered worse than death) Maximum: 1 (indicating full or perfect health)
Self-rated health | Baseline, 3 months and 6 months
  RESPONd participants will also be asked to complete the Euro Quality of Life (EuroQol) Visual Analog Scale (EQ-VAS) which assesses self-rated health on a vertical scale where respondents rate their overall health on the day of the survey.
  Range: 0 (worst imaginable health) to 100 (best imaginable health).
Rate of Emergency department (ED) visits | Baseline through study completion, an average of 18 months
  Frequency of ED usage rate per patient and per 1000
Rate of Hospital admissions | Baseline through study completion, an average of 18 months
  This will be measured by calculating number of inpatient stays per 1,000 people
Economic outcome measure - Incremental cost-effectiveness ratio (ICER) | Baseline through study completion, an average of 18 months
  The ICER ratio assesses cost-effectiveness and provides an estimate of the incremental cost for one additional unit of health outcome. To assess the effectiveness of the intervention, the ICER ratio per ED visit and hospital admission avoided will be applied to assess the number of visits avoided due to RESPONd. The number of ED visits and hospital admissions are also included as these are required to calculate the ICER ratio per visit type avoided.
Economic outcome measures - Quality adjusted life years (QUALYs) | Baseline through study completion, an average of 18 months
  Quality adjusted life years (QUALYs): A quality-adjusted life year is a summary measure used to evaluate the value of medical interventions in terms of the quality and quantity of life they produce. It combines both the duration of life and the health-related quality of life into a single index number. ICERs and net monetary benefit will be used to report QUALYs.

SECONDARY OUTCOMES:
Clinic outcome measure - Patient scheduling and clinic visit type | Baseline through study completion, an average of 18 months
  Information on the number, length, and type of visit (in-person or virtual; portal, telephone, email, or Zoom; Registered Nurse-led (RN-led) or Medical Oncologist-led (MO-led) will be obtained from the administrative database to assess clinical efficiency.
Clinic outcome measure - Number of patients that required additional intervention | Baseline through study completion, an average of 18 months
  The number of patients that required additional intervention after a clinic visit to determine if the triaged care was sufficient. The study nurse will also be required to keep track of the number of times needed to contact the medical oncologist (MO) address out of scope matters to also assess clinical efficiency.
Clinic outcome measure - Number of times the study nurse needed to contact the Medical Oncologist | Baseline through study completion, an average of 18 months
  The study nurse will keep track of the number of times needed to contact the Medical Oncologist (MO) to address out of scope matters to assess clinical efficiency.
Patient experience measure | At baseline, and 6 months/end of the intervention
  To understand patient perspectives, a web-based questionnaire will be disseminated to RESPONd participants via REDCap. Thirteen items on the patient experience measure are adapted from the Your Voice Matters patient-reported experience measure, developed by Cancer Care Ontario. Participants will be asked to rate each care experience using a three-point Likert scale:
  1. Yes, completely
  2. Yes, somewhat
  3. No.
  One question asks participants to measure the overall quality of all of their cancer care in the past 6 months using a five-point Likert scale:
  1. Poor
  2. Fair
  3. Good
  4. Very good
  5. Excellent
Staff experience measure | Quarterly - from baseline through study completion, an average of 18 months
  A researcher-developed web-based questionnaire designed to capture feedback from oncology clinic staff on the implementation and impact of the RESPONd program and the weekly team huddle.
  It includes questions on staff roles, clinic location, and perceived impacts on team collaboration, workflow efficiency, and the integration of patient data such as electronic PROs. The survey specifically evaluates how having access to weekly electronic PROs and participating in structured team huddles affects clinical decision-making and communication.
  Oncology clinic staff will be asked to rate each experience using a four-point Likert scale:
  1. Agree
  2. Somewhat Agree
  3. Somewhat disagree
  4. Disagree

CONTACTS AND LOCATIONS:
Overall Officials: Linda Watson, RN, PhD, Principal Investigator — Cancer Care Alberta, Alberta Health Services; Marni Armstrong, PhD, Study Director — Cancer Care Alberta, Alberta Health Services
Locations (4):
- Canada (4):
  - Arthur J. E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - High River Community Cancer Centre, High River, Alberta
  - Central Alberta Cancer Centre, Red Deer, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson L, Qi S, Link C, DeIure A, Afzal A, Barbera L. Patient-Reported Symptom Complexity and Acute Care Utilization Among Patients With Cancer: A Population-Based Study Using a Novel Symptom Complexity Algorithm and Observational Data. J Natl Compr Canc Netw. 2023 Feb;21(2):173-180. doi: 10.6004/jnccn.2022.7087. PMID 36791760